CLINICAL TRIAL: NCT03101930
Title: Cardiovascular Effects of GLP-1 Receptor Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, James Matt Luther, Associate Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB# 170213
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Obesity; PreDiabetes
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Liraglutide; Sitagliptin Phosphate; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment with liraglutide or sitagliptin will be masked using matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- liraglutide (Experimental): Subjects in the liraglutide group will receive subcutaneous liraglutide (0.6 mg/d for one week, 1.2 mg/d for one week, and then 1.8 mg/d for 12 weeks) and oral placebo.
  Interventions: Drug: Liraglutide; Drug: Placebos; Drug: Exendin (9-39)
- sitagliptin (Active Comparator): Subjects in the sitagliptin group will receive subcutaneous placebo daily and sitagliptin 100 mg/d orally for 14 weeks.
  Interventions: Drug: Sitagliptin; Drug: Placebos; Drug: Exendin (9-39)
- hypocaloric diet (Active Comparator): Subjects in the hypocaloric diet group will be given a caloric goal designed to achieve a weight loss similar to that expected in the liraglutide treatment arm based on his or her resting energy expenditure. Subjects will be provided counseling and written instructions on how to achieve their daily caloric goal, including use of their own mobile phone applications to monitor caloric intake. To assure compliance with the prescribed caloric goal, subjects will meet with the study dietitian every other week for problem solving and review of diet intake logs.
  Interventions: Other: hypocaloric diet; Drug: Placebos; Drug: Exendin (9-39)

INTERVENTIONS:
Drug: Liraglutide — subcutaneous liraglutide daily
  Arms: liraglutide
Drug: Sitagliptin — oral sitagliptin daily
  Arms: sitagliptin
Other: hypocaloric diet — Reduced calorie intake to achieve weight loss.
  Arms: hypocaloric diet
Drug: Placebos — Subjects in the liraglutide arm will receive a placebo for sitagliptin. Those in the sitagliptin arm will receive a placebo for liraglutide. All subjects will receive a placebo for Exendin 9-39.
Drug: Exendin (9-39) — All subjects will receive Exendin (9-39) or matching placebo in crossover fashion during study days on the first and third days of the second week after randomization and again on the 5th and 7th days of the 14th week of treatment.

SUMMARY:
This project tests the principle hypothesis that stable glucagon like peptide-1 (GLP-1) analogues have specific GLP1R-dependent beneficial effects on vascular endothelial function, fibrinolysis and inflammation in obesity that exceed the benefits of weight loss, and that genetic or other individual factors that modulate GLP1R sensitivity can modify the effect of these analogues on cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women,
2. Age 18 to 65 years, and
3. FPG (100-125 mg/dL) or, IGT (two-hour plasma glucose 140-199 mg/dL) or, HbA1C 5.7-6.4%
4. BMI≥30 kg/M2
5. The ability to provide informed consent before any trial-related activities.

Exclusion Criteria:

1. Diabetes type 1 or type 2, as defined by a FPG of 126 mg/dL or greater, a two-hour plasma glucose of 200 mg/dL or greater, or the use of anti-diabetic medication
2. Resistant hypertension, defined as hypertension requiring the administration of more than three anti-hypertensive agents including a diuretic to achieve control
3. Use of spironolactone
4. Known or suspected allergy to trial medications, excipients, or related products.
5. Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma
6. Personal history of non-familial medullary thyroid carcinoma
7. History of pancreatitis
8. Contraindications to study medications, worded specifically as stated in the product's prescribing information
9. Pregnancy or breast-feeding. Women of child-bearing potential will be required to have undergone tubal ligation or to be using an oral contraceptive or barrier methods of birth control
10. Subjects who have participated in a weight-reduction program during the last six month or whose weight has increased or decreased more than two kg over the preceding six months
11. Cardiovascular disease such as myocardial infarction within six months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
12. Treatment with anticoagulants
13. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
14. History or presence of immunological or hematological disorders
15. Diagnosis of asthma requiring regular inhaler use
16. Clinically significant gastrointestinal impairment that could interfere with drug absorption
17. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >3.0 x upper limit of normal range)
18. Individuals with an eGFR<30 mL/min/1.73 m2 or with a UACR >1000µg/mg, where eGFR is determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine is expressed in mg/dL and age in years: eGFR (mL/min/1.73m2)=186 • Scr-1.154 • age-0.203 • (1.212 if black) • (0.742 if female)
19. Hematocrit <35%
20. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
21. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
22. Treatment with lithium salts
23. History of alcohol or drug abuse
24. Treatment with any investigational drug in the one month preceding the study
25. Previous randomization in this trial
26. Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
27. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M. Luther, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.

REFERENCES:
- See also: Study Pre-print on medRxiv — https://www.medrxiv.org/content/10.1101/2022.02.23.22271434v1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: CONSORT flow details:
  * 329 signed consent.
  * 178 individuals did not meet inclusion/exclusion criteria.
  * 35 individuals declined to participate.
  * 23 individuals did not return for subsequent visits.
  * 93 individuals randomized.
  * 88 individuals completed study days.
Period: Overall Study
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Started | 46 | 23 | 24
Completed | 44 | 22 | 22
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet | Total
Number analyzed (Participants) | 46 | 23 | 24 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (9.9) | 52.8 (10.5) | 48.9 (12.1) | 50.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 16 | 14 | 63
  Male | 13 | 7 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 44 | 21 | 23 | 88
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 4 | 13
  White | 38 | 18 | 19 | 75
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 23 | 24 | 93
Flow mediated dilation [Mean (Standard Deviation); unit: Percentage] — Population: Due to missed study visits and missing samples, there is incomplete data for the following arms/time periods: Liraglutide 4, Sitaglipin 1, Hypocaloric Diet 3
  Percentage
    number analyzed (Participants) | 42 | 22 | 21 | 85
    (all) | 10.5 (5.2) | 10.4 (5.37) | 10.2 (5.3) | 10.4 (5.2)
Urine Albumin-Creatinine ratio [Mean (Standard Deviation); unit: mg/g] — mg albumin/g creatinine Population: Participants who were randomized to intervention but did not complete study day measurements are not included: Liraglutide 2, Sitagliptin 1, Hypocaloric Diet 2
  mg/g
    number analyzed (Participants) | 44 | 22 | 22 | 88
    (all) | 12.04 (23.6) | 7.85 (7.6) | 6.3 (3.8) | 9.6 (17.3)
Plasminogen Activator Inhibitor-1, plasma [Mean (Standard Deviation); unit: U/mL] — plasma PAI-1 (U/mL) Population: Due to missed study visits and missing samples, there is incomplete data for the following arms/time periods: Liraglutide 3, Sitaglipin 2, Hypocaloric Diet 4
  U/mL
    number analyzed (Participants) | 43 | 21 | 20 | 84
    (all) | 20.2 (9.2) | 18.5 (8.6) | 18.5 (8.0) | 19.4 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation
Description: Brachial artery diameter is measured under basal conditions and during reactive hyperemia (Flow Mediated Dilation as %)
Time Frame: Baseline to 2 and 14 weeks
Population: Incomplete data due to missed study visits and missing samples in the following time periods/arms (n= number of participants with missing data):
  * Liraglutide/Placebo: Week 2 (n=5); Week 14 (n=4)
  * Liraglutide/Exendin: Week 2 (n=11); Week 14 (n=12)
  * Sitagliptin/Placebo: Week 2 (n=2)
  * Sitagliptin/Exendin: Week 2 (n=3); Week 14 (n=2)
  * Diet/Placebo: Week 2 (n=1); Week 14 (n=6)
  * Diet/Exendin: Week 2 (n=7); Week 14 (n=11)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
Percentage
  Baseline to 2 weeks (Placebo infusion): number analyzed (Participants) | 39 | 20 | 21
  Baseline to 2 weeks (Placebo infusion) | 0.71 (4.82) | 2.06 (6.42) | 1.24 (5.09)
  Baseline to 2 weeks (Exendin infusion): number analyzed (Participants) | 33 | 19 | 15
  Baseline to 2 weeks (Exendin infusion) | 0.48 (5.81) | 0.13 (4.49) | 1.43 (7.09)
  Baseline to 14 weeks (Placebo infusion): number analyzed (Participants) | 40 | 22 | 16
  Baseline to 14 weeks (Placebo infusion) | 1.43 (5.33) | 1.59 (5.74) | 1.01 (5.38)
  Baseline to 14 weeks (Exendin infusion): number analyzed (Participants) | 32 | 20 | 11
  Baseline to 14 weeks (Exendin infusion) | 1.73 (5.22) | 1.42 (5.88) | 0.42 (4.28)

2. Primary Outcome: Urine Albumin-to-creatinine Ratio
Description: Ratio of urine albumin to creatinine in a spot urine collected after overnight rest
Time Frame: Baseline to 13 weeks
Population: Due to missed study visits and missing samples, there is incomplete data for the following arms/time periods:
  Liraglutide: 2 participants; Diet: 6 participants
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
mg/g
  Baseline | 12.0 (23.6) | 7.9 (7.6) | 6.3 (3.8)
  13 Weeks: number analyzed (Participants) | 42 | 22 | 16
  13 Weeks | 10.5 (14.8) | 9.2 (10.7) | 10.1 (19.4)

3. Primary Outcome: Change in Plasminogen Activator Inhibitor-1
Description: Plasma plasminogen activator inhibitor-1 antigen
Time Frame: Baseline to 2 and 14 weeks
Population: Due to missed study visits and missing samples, there is incomplete data for the following arms/time periods:
  Liraglutide: Baseline: 2 participants/Week 14: 3 participants; Sitagliptin: Baseline: 1 participants/Week 14: 1 participants; Diet: Baseline: 3 participants/Week 14: 6 participants
Measure: Mean (Standard Deviation); unit: units/mL
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
units/mL
  Baseline to 2 weeks: number analyzed (Participants) | 42 | 21 | 19
  Baseline to 2 weeks | -2.4 (7.8) | -1.3 (8.3) | 1.1 (6.9)
  Baseline to 14 weeks: number analyzed (Participants) | 41 | 21 | 16
  Baseline to 14 weeks | -3.7 (8.7) | 1.3 (6.3) | -3.6 (6.6)

4. Secondary Outcome: Blood Pressure
Description: The mean of three systolic blood pressure measurements one minute apart using a oscillometric recording device with patient in supine position
Time Frame: Baseline, and after 2 weeks and 14 weeks of treatment
Population: Due to missed study visits there is incomplete data for the following arms/time periods:
  Liraglutide 14 weeks- 2 participants; Diet 14 weeks: 5 participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
mmHg
  Baseline | 124.1 (7.7) | 120.2 (11.3) | 127.7 (8.3)
  2 weeks | 122.9 (6.3) | 117.5 (11.3) | 121.7 (6.8)
  14 weeks: number analyzed (Participants) | 42 | 22 | 17
  14 weeks | 122.2 (7.8) | 118.2 (13.9) | 119.7 (11.1)

5. Secondary Outcome: Heart Rate
Description: The mean of three measurements with the patient in the supine position
Time Frame: Baseline, and after 2 weeks and 14 weeks of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
Beats per minute
  Baseline | 64.9 (7.5) | 67.2 (9.0) | 63.8 (8.8)
  2 weeks | 68.9 (6.4) | 66.2 (9.2) | 63.2 (9.5)
  14 weeks: number analyzed (Participants) | 42 | 22 | 17
  14 weeks | 68.9 (5.6) | 65.9 (8.5) | 61.7 (7.9)

6. Secondary Outcome: Fasting Glucose
Description: Blood glucose collected after overnight fast
Time Frame: Baseline, and after 2 weeks and 14 weeks of treatment
Population: Due to missed study visits there is incomplete data for the following arms/time periods:
  Liraglutide Baseline-1, 2 weeks 1, 14 weeks- 2 participants; Sitagliptin 2 weeks 1, 14 weeks- 1 participants; Diet 14 weeks: 5 participants
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
mg/dl
  Baseline: number analyzed (Participants) | 43 | 22 | 22
  Baseline | 95.3 (8.6) | 97.6 (10.0) | 94.5 (12.0)
  2 weeks: number analyzed (Participants) | 43 | 21 | 22
  2 weeks | 84.26 (7.9) | 93.9 (8.1) | 92.4 (11.3)
  14 weeks: number analyzed (Participants) | 42 | 21 | 17
  14 weeks | 85.2 (7.3) | 96.6 (5.6) | 91.2 (9.8)

7. Secondary Outcome: Fasting Insulin
Description: Plasma insulin collected after overnight fast
Time Frame: Baseline, and after 2 weeks and 14 weeks of treatment
Population: Due to missed study visits or missing data there is incomplete data for the following arms/time periods:
  Liraglutide 2 weeks 3, 14 weeks- 3 participants; Sitagliptin 2 weeks 2, 14 weeks- 1 participants; Diet 14 weeks: 5 participants
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 44 | 22 | 22
uU/mL
  Baseline | 22.7 (16.8) | 23.3 (14.4) | 26.7 (21.2)
  2 weeks: number analyzed (Participants) | 41 | 20 | 22
  2 weeks | 18.3 (12.5) | 29.4 (25.4) | 19.7 (16.5)
  14 weeks: number analyzed (Participants) | 41 | 21 | 17
  14 weeks | 20.3 (14.7) | 26.0 (19.0) | 20.3 (13.7)

8. Other Pre Specified Outcome: Change in Weight
Description: Weight measured in light clothing without shoes
Time Frame: Change from baseline to 14 weeks
Population: Due to missed study visits or missing data there is incomplete data for the following arms/time periods:
  Liraglutide 2 participants; Diet 5 participants
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
Number analyzed (Participants) | 42 | 22 | 17
kg | -2.72 (3.44) | -0.71 (2.12) | -4.95 (3.98)

ADVERSE EVENTS:
Time Frame: After randomization to 14 weeks
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time of randomization through participant completion at each screening visit, study day, and at week 4, week 8 and week 12 check-ins.
Arm/Group | Liraglutide | Sitagliptin | Hypocaloric Diet
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/46 | 1/23 | 1/24
Other Adverse Events (participants affected / at risk) | 26/46 | 6/23 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=46) | Sitagliptin (N=23) | Hypocaloric Diet (N=24)
Cellulitis/abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis and hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=46) | Sitagliptin (N=23) | Hypocaloric Diet (N=24)
Nausea (Gastrointestinal disorders) | 8 (8) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Study day procedure adverse event (Surgical and medical procedures) | 22 (41) | 6 (9) | 6 (9) — Including nausea or abdominal pain from mixed meal tolerance test, pain from ultrasound flow-mediated dilation technique or from subcutaneous adipose tissue liposuction, headache from nitroglycerin administration.
Injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Lightheaded (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study enrollment and conduct interrupted due to COVID-19 pandemic. Exendin not available for all study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03101930/Prot_SAP_000.pdf